CLINICAL TRIAL: NCT07214987
Title: A Phase 2 Study of Toripalimab in Combination With Cisplatin and Docetaxel (PDT) for Induction Therapy in CPS-Positive Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: PDT For Induction Therapy For Head And Neck Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Coherus Oncology, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas J. Roberts, MD, Principle Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-494
Record Dates: First submitted 2025-09-25; First posted 2025-10-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma; Head and Neck Cancer Squamous Cell Carcinoma; Head and Neck Cancer
Keywords: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PDT (cisplatin + docetaxel + toripalimab) induction therapy (Experimental): Toripalimab, cisplatin, and docetaxel will be given once every 21 days, +/- a window of 5 days, by intravenous infusion. On day 1 of each cycle, the pre-determined dose of toripalimab will be administered over about 60 minutes. The pre-determined dose of docetaxel will then be administered over about 1 hour. After docetaxel, the pre-determined dose of cisplatin will be administered over about 1-3 hours. This will continue for up to 3 cycles. Participants may be pre-medicated with drugs to reduce the chance of having a sensitivity reaction to the study treatment. The decision to pursue definitive chemoradiotherapy should be made by a multidisciplinary team specializing in treating head and neck cancers. For patients receiving chemoradiotherapy, the recommended concurrent chemotherapy regimen used with radiotherapy is weekly cisplatin.
  Interventions: Drug: Toripalimab-tpzi; Drug: Cisplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Toripalimab-tpzi — Toripalimab-tpzi is a humanized IgG4 monoclonal antibody specific against human PD-1.
  Other Names: JS001; TAB001; CHS-007; LOQTORZI
Drug: Cisplatin — Cisplatin is an injectable chemotherapy agent classified as a platinum-based alkylating agent.
Drug: Docetaxel — Docetaxel is a taxane chemotherapy agent.

SUMMARY:
This research study is being done to assess the safety and tolerability of toripalimab in combination with cisplatin and docetaxel (PDT) induction therapy for patients with CPS-positive locally advanced head and neck squamous cell carcinoma (HNSCC).

DETAILED DESCRIPTION:
This is a single arm phase II study to assess treatment-related adverse events (TRAEs) and efficacy of PDT. The study employs a Simon two-stage design. After 12 evaluable participants start treatment with at least 2 participants experiencing no grade 3 or higher TRAEs during induction therapy, then enrollment will continue to the target number of participants of 26. Participants will receive treatment for three cycles or until disease progression, they experience unacceptable side effects, their condition changes rendering them unacceptable for further treatment, or they withdraw from the study. Participants will be followed for two years from registration. Coherus Biosciences, Inc. is supporting this research study by providing the study drug, toripalimab, and funding for research activities. The U.S. FDA has not approved toripalimab for CPS-positive locally advanced HNSCC but has approved it for other forms of head and neck cancer. Toripalimab is a lab-made antibody that works by allowed the immune system to attack cancer cells more effectively. Toripalimab is currently sold as LOQTORZI and is used with cisplatin and gemcitabine to treat nasopharyngeal carcinoma. The U.S. FDA has approved cisplatin and docetaxel as a treatment option for multiple types of cancers, including head and neck small cell carcinoma. Cisplatin is a chemotherapy agent that works by binding to cancer cells and initiating cell death. Docetaxel is a chemotherapy agent made from a compound found in the European yew tree. Docetaxel works by stabilizing tiny structures within cancer cells, prevent cell growth and, ultimately leading to cell death. The combination of toripalimab with cisplatin and docetaxel for induction therapy is investigational.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a new diagnosis of histologically or cytologically confirmed squamous cell carcinoma (SCC) of the oral cavity, oropharynx, hypopharynx, larynx, nasopharynx, sinonasal cavities or unknown primary HNSCC.
* Participants with HPV-independent SCC or HNSCC or other head and neck subsites must have stage III or non-metastatic stage IV at the time of diagnosis. Participants with HPV-associated oropharynx SCC must have stage II or stage III disease.
* Participants must be determined by the investigator to be candidates for induction systemic therapy due to reasons such as the extent of primary tumor at the time of diagnosis, rate of progression, symptom burden or potential benefit of cytoreduction prior to definitive local therapy.
* CPS ≥ 1%
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of toripalimab in combination with cisplatin and docetaxel in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status ≤ 1
* Life expectancy of greater than 12 weeks.
* Participants must meet the following organ and marrow function as defined below:

Hemoglobin ≥8.0 g/dL absolute neutrophil count ≥1500/mcL platelets ≥100,000/mcL total bilirubin ≤ 2 institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤ 2 × institutional ULN creatinine ≤ 2 x institutional ULN OR glomerular filtration rate (GFR) ≥ 45 mL/min/1.73 m2

* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Because immunotherapy agents as well as cisplatin and docetaxel are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of toripalimab administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Diagnosis of EBV-associated nasopharynx squamous cell carcinoma
* Strong clinical suspicion or histologic confirmation of cutaneous squamous cell carcinoma
* Histology other than squamous cell carcinoma.
* Proven distant metastases (below the clavicle) by clinical or radiographic measures.
* Prior radiotherapy to the head and/or neck with the exception of radiation for cutaneous malignancies involving radiation fields that do not overlap with areas of current disease involvement.
* Pre-existing peripheral neuropathy CTCAE grade 2 or higher
* Participants who are receiving any other investigational agents for this condition.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to toripalimab, cisplatin or docetaxel.
* An autoimmune condition requiring treatment with systemic corticosteroids within the past 30 days. Long-term steroid replacement for patients with adrenal insufficiency is allowed.
* Any second malignancy that required antineoplastic therapy in the previous 6 months.
* Participants receiving any medications or substances that are moderate or strong inhibitors or inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product.
* Pregnant women are excluded from this study because toripalimab, cisplatin and docetaxel have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with toripalimab, cisplatin and docetaxel, breastfeeding should be discontinued if the mother is treated with toripalimab. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-03-09 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion Grade 3-5 TRAE-free during induction therapy | Day 1 of Cycle 1 (each cycle is 21 days) to Day 10 of Cycle 3 (end of induction therapy).
  Assessed using NCI Common Terminology for Adverse Event (CTCAE) version 5.0. The rate of patients with grade 3+ TRAEs-free during induction therapy will be summarized as a proportion with a corresponding exact 95% confidence interval (CI) (if the trial closes to accrual after the first stage), or a proportion with a corresponding 95% two-stage confidence interval (CI) if the trial closes to accrual after the second stage.

SECONDARY OUTCOMES:
Proportion Grade 3-5 TRAE-free during curative-intent treatment | Day 1 of Cycle 1 (each cycle is 21 days) through the completion of 7 weeks of definitive chemoRT or 30 days after surgery for patients who undergo surgery and are deemed by the treating team to not require additional post-operative therapy.
  Assessed using NCI Common Terminology for Adverse Event (CTCAE) version 5.0. The rate of participants grade 3+ TRAEs-free during the entire period of curative-intent treatment will be summarized as a proportion with a corresponding exact 95% confidence interval (CI) (if the trial closes to accrual after the first stage), or a proportion with a corresponding 95% two-stage confidence interval (CI) if the trial closes to accrual after the second stage.
Overall Response Rate (ORR) after PDT induction therapy | Day 1 of Cycle 1 (each cycle is 21 days) to day 1 of cycle 3.
  The overall response rate (ORR) will be summarized as a proportion with a corresponding exact 95% two-stage confidence interval (CI).
Overall Response Rate (ORR) after curative-intent therapy | Day 1 of Cycle 3 (each cycle is 21 days) to day of 3-month follow-up visit.
  The overall response rate (ORR) will be summarized as a proportion with a corresponding exact 95% two-stage confidence interval (CI).
Event-free Survival | Day 1 of Cycle 1 (each cycle is 21 days) to date of death or for up to 2 years from study registration (whichever comes first).
  The Kaplan-Meier method will be used to estimate time-to-event endpoints with corresponding 95% confidence intervals (CIs) for the median or time-specific event time.
Overall Survival | Day 1 of Cycle 1 (each cycle is 21 days) to date of death or for up to 2 years from study registration (whichever comes first).
  Overall survival is the time from start of treatment to death due to any cause. The Kaplan-Meier method will be used to estimate time-to-event endpoints with corresponding 95% confidence intervals (CIs) for the median or time-specific event time.
Participant's Quality of Life | Baseline until to 2 years from study registration.
  Patient-Reported Outcomes Measurement Information System Global 10 (PROMIS-10) Physical Health T-score and Global Mental Health T-score will be summarized descriptively via PROMIS-10 scores. The minimum score is 16 and the maximum is 68. A higher score is associated with better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Roberts, MD, MBA, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Thomas Roberts, MD, MBA at 617-726-5130. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation